CLINICAL TRIAL: NCT03312829
Title: Team Sepsis: Fast I(n)Dentification of PATHogens (FINDPATH)
Brief Title: FINDpath: Fast I(n)Dentification of PATHogens
Acronym: FINDpath
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: FINDpath14
Record Dates: First submitted 2014-08-29; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Respiratory Tract Infections; Critical Illness
MeSH Terms: conditions — Respiratory Tract Infections; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dr. Surette's laboratory has optimized methods or enrichment of bacterial cells directly from blood allowing for bacterial nucleic acid isolation suitable for molecular profiling with as little as 1ml of blood. However, this methodology does have a limitation in that the detection of bacterial DNA does not necessarily imply that there are corresponding viable bacterial present.
  To overcome the lack of accuracy of this method, the investigators propose to apply our optimized methods for bacterial cell enrichment from blood and nucleic acid isolation to ribosomal RNA rather than DNA.
Oversight: Data Monitoring Committee: No

SUMMARY:
Sepsis is the body-wide response to infection. People who develop sepsis have an increased risk of dying. One of the greatest challenges in sepsis is determining what is the pathogen (bacteria or virus for example) in a timely manner so the most specific antibiotics can be given to treat the infection. Patients presenting to the hospital and the intensive care unit often have lung infections. In this study the investigators plan to develop new techniques to rapidly (less than 6 hours) identify bacteria growing in the airways of patients on ventilators. The investigators will obtain these samples by suctioning the airways (a routine procedure) and comparing the bacterial cultures grown by novel culture media with the usual techniques in the hospital microbiology laboratory. At the same time the investigators will collect a blood sample. This blood sample will be used to isolate the bacterial genetic material and use this to compare with bacteria grown on the culture media from the clinical and the research laboratory. The investigators will also collect information on the patient's course in hospital. These pilot study results will allow us to integrate this new technique into routine patient care.

DETAILED DESCRIPTION:
The trial design is a pilot observational feasibility study within three intensive care units at the Hamilton General Hospital, which is composed of both medical and surgical patient populations where waived consent has been confirmed and approved by the Hamilton Integrated Research Ethics Board. The study sample will include 50 patients over the age of 16 that will be mechanically ventilated for greater than 48 hours with no antibiotic use for the past 24 hours and meet the Johanson Criteria for Ventilator Associated Pneumonia (VAP) as the gold standard for diagnosis still remain controversial. This Johanson criteria maintains patients must have 2 out of three criteria to be enrolled in the study and that criteria includes either a leukocyte count >12,000/mm³ , Fever >38.0ºC and/or a new onset of purulent endotracheal secretions or change in the character of sputum. Chest x-rays for examination of a new or progressing infiltrate will be assessed but will not be used for initial inclusion criteria but possibly in the conclusions when attempting to differentiate VAP from VAT.

Recruitment of eligible patients maintains the need for daily screening of patients which will be done primarily by myself as the co-investigator and from a research assistant through the secure hospital patient data system. However education of the frontline staff particularly nursing, respiratory therapists, physiotherapists and staff physicians who will have direct contact with potential subject is also essential for successful recruitment, coordination and timing of enrollment. I will create and hold education sessions for all frontline staff outlining the purpose of the study, patient enrollment criterion and proper sample collection procedures as well as continual bedside education throughout the course of the study to ensure all staff will have the information to identify potential study patients.

Once patients are identified as meeting criteria for enrollment, the research assistant will be notified at which time the frontline staff will retrieved a premade package for the sample collection. Using a sterile catheter and a clean technique, two separate tracheal aspirates will be acquired from the subject and placed in their specialized clinical or research sputum trap. To acquire two samples, sterile saline irrigation will be permitted and if needed the splitting of the specimen into the separated collection traps. Concurrently a tube of blood as well as one set of blood cultures from an established indwelling access (either central line, arterial line or peripheral blood draw) will be drawn. Clinical lab labels will be placed on one sputum sample and the set of blood cultures and sent routinely to the microbiology lab. The research lab bag will contain the second sputum sample and blood tube labelled with patient identification number and the time of sample collection. To ensure the ability of culturing for anaerobic bacteria in the research laboratory, an anaerobic pack will be placed in the research sample bag with the sputum sample and blood tube as well as a damp paper towel. The sample bag will then be voided of air and sealed. The research bag is labelled as well with patient identification number and date/time of sample collection which is then sent to the clinical microbiology lab. The clinical laboratory is then notified of the incoming research sample which will need to be transported to the research laboratory via established laboratory transportation protocols. Once the sample is sent, the co-investigator is notified again and clinical data (leukocytes, hemoglobin, platelets, arterial blood gases, temperature, Glasgow coma scale, oxygen requirements, high/low respiratory rate, heart rate, and blood pressure) for the day of collection and for the following six days including complete ICU antibiotic usage, extubation date and final patient outcome after 30 days can be collected and entered into a secure RedCap database. Communication to the research laboratory will be the responsibility of the co-investigator to ensure samples have arrived and can be plated in the time set out within the study protocol. Transportation of the samples are available from 0700 until 2000 Monday through Sunday so identification of potential enrollment , and collection of samples will be encouraged during these times to ensure successful arrival and processing of samples at the research laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 16yrs
2. ICU patients at the General site with a suspected tracheobronchitis or VAP
3. Ventilated for greater than 48 hours
4. No antibiotics for 24 hours prior to collection of specimens

Exclusion Criteria:

1. Hopeless prognosis
2. Have received antibiotics 24 hours prior to collection of specimens
3. Previously enrolled in FINDPATH

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult Intubated ICU Patients
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of eligible patients recruited by front line respiratory and nursing staff | 12 months
  Staff identify and enrolled 80% of eligible patients

SECONDARY OUTCOMES:
Correlation between clinical lab and research laboratory for pathogen identification | 18 months
  What pathogens are identified by the research lab that are not cultured in the clinical laboratory

OTHER OUTCOMES:
Number of patients with ventilator specific outcomes according to Ventilator Associated Pneumonia guidelines | 24 months
  Morbidity and Mortality at 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Alison Fox-Robichaud, MD, Principal Investigator — Hamilton Health Sciences; McMaster University; Stephanie Rotella, BSc, RRT, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences - General Site, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
analysis in progress